CLINICAL TRIAL: NCT03639103
Title: Medium-Long-Term Clinical and Radiographic Outcomes of Minimally Invasive Distal Metatarsal Metaphyseal Osteotomy for Central Primary Metatarsalgia and Predictive Value of Maestro Criteria
Brief Title: Clinical and Radiographic Outcomes of Distal Metatarsal Metaphyseal Osteotomy for Central Primary Metatarsalgia
Acronym: DMMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Carlo Biz, Orthopedic surgeon, Assistant Professor, University of Padova
Other Study IDs: 4064/AO/17
Record Dates: First submitted 2018-07-31; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Metatarsalgia Bilateral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Distal Metatarsal Metaphyseal Osteotomy (DMMO) — The scalpel is advanced at an oblique angle of about 45° until it reaches the dorsal aspect of the distal metatarsal bone to undergo osteotomy. First a bone rasp specific for percutaneous surgery is used to separate the periosteum at the level of the osteotomy site. A Shannon Isham burr is introduced until it reaches the metatarsal neck where the periosteum was previously removed. Fluoroscopy is used to confirm the correct position of the osteotomy site. The lateral cortical surface is cut first, then the plantar, medial, and lastly, the dorsal cortical surface. During the osteotomy process, the incision site is irrigated by normal saline, as the burr can cause excessive heat, causing skin burn and resulting subsequently in fibrosis and pseudoarthrosis at the bone level.
  Other Names: DMMO PERCUTANEOUS SURGERY

SUMMARY:
The primary propose of this prospective study is to specifically evaluate the safety and effectiveness of Minimally Invasive Distal Metatarsal Metaphyseal Osteotomy (DMMO) in treating patients with persistent central primary metatarsalgia, associated or not to hallux valgus and lesser toe deformities, identifying possible contraindications in relation to some demographic parameters (age, gender, BMI, and smoking). The second objective is to verify the potential of DMMO in restoring a harmonious foot morphotype according to Maestro's criteria and if these radiographic parameters are correlated with clinical outcomes, maintaining the predictive value of these criteria during preoperative planning also for this percutaneous surgery.

DETAILED DESCRIPTION:
A consecutive series of patients with metatarsalgia is consecutively enrolled and treated by DMMO. According to Maestro criteria, pre-operative planning is carried out by both clinical and radiological assessment. Patient demographic data, AOFAS scores, 17-Foot Functional Index, Manchester-Oxford Foot Questionnaire, SF-36, VAS, and complications are recorded. Maestro parameters, relative morphotypes, and bone callus formation are assessed. Statistical analysis is carried out (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* forefoot persistent pain;
* presence or not of forefoot plantar hyperkeratosis lesions;
* ineffective conservative and orthotic treatment performed for at least 6 months.

Exclusion Criteria:

* arthritis and stiffness of MTP joint;
* congenital deformities of the foot;
* hallux rigidus;
* Freiberg infraction;
* Morton's neuroma;
* diagnosis of rheumatic, metabolic, neurologic, infective, or psychiatric pathologies;
* previous trauma;
* foot and ankle surgery,
* any form of secondary or iatrogenic metatarsalgia.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of central primary metatarsalgia between M2 and M4 of a biomechanical etiology in the plantar foot area are enrolled consecutively and prospectively with precise inclusion criteria. Ages range from 18 to 90 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the 100-point hallux metatarsophalangeal-interphalangeal scale (AOFAS) changes | preoperatively, 3-, 6-, 12-months
  The AOFAS score includes 9 questions related to pain, function and alignment; a score of 90-100 is considered excellent; 75-89 as good; 50-74 as fair and less than 49 points is considered a failure or a poor outcome.
Evaluation of the Foot Functional Index changes | preoperatively, 3-, 6-, 12-months
  The Foot Functional Index to measure the persistence of pain, disability, and restriction of activity with 17 number rating scales from 0 to 10. The maximum score is 100, which indicates complete disability.
Evalutation of the Manchester-Oxford Foot Questionnaire changes | preoperatively, 3-, 6-, 12-months
  The Manchester-Oxford Foot Questionnaire to establish how frequent the restrictions in specific situations were, including 16 questions divided into three basic domains: pain (five), walking/standing (seven), and social interaction (four). Scores for each domain are calculated by summing the responses to each item within a given domain. Raw scores can be converted to a 0-100 metric where 100=most severe.

SECONDARY OUTCOMES:
Radiographic classification according to Maestro and Besse criteria | before surgery, at one-month after surgery and at different follow-ups (3-, 6-, 12-month, and last)
  Our sample is classified radiographically according to Maestro and Besse criteria, adding to this classification one more group to include those feet that did not reflect any morphotype as defined by Maestro parameters. The radiographic evaluations includes the Maestro criteria index using the preoperative and the last follow up. The relative length of each metatarsal is determined by drawing a line perpendicular to the axis of the foot and then measuring the distances (in millimeters) from each metatarsal head to this line , while also taking into account the relationship between the length of metatarsal M1 and the length of the remaining metatarsal bones.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Biz, MD, Principal Investigator — Padua University Orthopaedic Clinic
Locations (1):
- Padua Univeristy Orthopaedic Clinic, Padua, Italy

IPD SHARING:
Plan to Share IPD: No